CLINICAL TRIAL: NCT01154205
Title: Sheba Medical Center Home Monitoring Clinic Registry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. David Luria, Heart Center at Sheba Medical Center
Other Study IDs: SHEBA-09-7598-DL-CTIL
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Clinical Workload Assessment Based Upon a Home Monitoring System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients post implantation of ICD or CRTD

SUMMARY:
The purpose of the registry is to assess workload of a Home Monitoring based follow up for Biotronik ICD and CRTD patients.

ELIGIBILITY:
Inclusion Criteria:

* Approved indication for ICD or CRTD
* Implanted with or replaced with a Biotronik Lumax device
* Patient willing and able to sign consent form
* Willing and able to attend clinic visits and follow up schedule
* Transmission of more than 80% at 3-month follow up
* Patient older than 18 years

Exclusion Criteria:

* no indication for ICD or CRTD implant
* Life expectancy shorter than 12 months
* Pregnancy
* Participation in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with an ICD or CRTD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-06; Study Completion 2012-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Ramat Gan, Israel